CLINICAL TRIAL: NCT01300403
Title: Acute Physiological Effects of Expiration With the Glottis Open in Lateral Posture (ELTGOL) and Flutter Valve in Dynamic and Static Pulmonary Volumes of Patients With Bronchiectasis
Brief Title: Physiological Effects of Expiration With the Glottis Open in Lateral Posture (ELTGOL) and Flutter Valve in Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Centro Universitário Augusto Motta (Other)
Responsible Party: Fernando Silva Guimarães, Augusto Motta University Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02/2009
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2010-09

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Exhalation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- FLUTTER (Experimental): Since this was a crossover study, all patients performed all interventions in a randomized order.
  Interventions: Other: Flutter valve
- ELTGOL (Experimental): Since this was a crossover study, all patients performed all interventions in a randomized order.
  Interventions: Other: expiration with the glottis open in lateral posture (ELTGOL)
- CONTROL (Active Comparator): Since this was a crossover study, all patients performed all interventions in a randomized order.
  Interventions: Other: Control

INTERVENTIONS:
Other: Flutter valve — Flutter valve is a physiotherapy device commonly used for the treatment of pulmonary hypersecretive conditions. The patients is taught to exhale through the device, producing positive expiratory pressure and flow oscillations. In this study the intervention took 15 minutes. During this period the patients were free to cough.
  Arms: FLUTTER
Other: expiration with the glottis open in lateral posture (ELTGOL) — This technique is a maneuver of slow expiration with the glottis open, with the subject in lateral posture. The patients performed three sets of 10 repetitions in left and right lateral decubitus.
  Arms: ELTGOL
Other: Control — Patients were instructed to stay comfortably seated during 15 minutes. After this period they were stimulated to cough during a five minutes period.
  Arms: CONTROL

SUMMARY:
This study aimed to evaluate the acute physiological effects of expiration with the glottis open in lateral posture (ELTGOL) and Flutter valve in dynamic and static lung volumes in patients with bronchiectasis and, secondarily, to study the effect of these techniques in sputum production.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinical and radiological criteria of bronchiectasis

Exclusion Criteria:

* heart failure
* pneumonia
* chest pain
* inability to perform the procedures
* asthma
* cystic fibrosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Dynamic and static lung volumes | In the week 1, 2 and 3. Before (baseline) and after each intervention.
  Dynamic and static lung volumes were assessed by forced spirometry and plethysmography.

SECONDARY OUTCOMES:
Sputum production | Sputum was colected during the interventions
  The expectorated secretions were collected using a sputum trap and quantificated by its dry weight.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando S Guimarães, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Universitário Pedro Ernesto, Rio de Janeiro, Rio de Janeiro, Brazil